CLINICAL TRIAL: NCT03765476
Title: Validation of a Computer-based Training Program for Patients With Alcohol Use Disorder
Brief Title: Validation of a Training Program for Patients With Alcohol Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SALIENCE
Record Dates: First submitted 2018-10-23; First posted 2018-12-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: one group receives add-on- intervention "SALIENCE"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU (Active Comparator): treatment as usual
  Interventions: Behavioral: TAU
- TAU plus SALIENCE (Experimental): treatment as usual plus computer-based intervention "SALIENCE"
  Interventions: Behavioral: SALIENCE; Behavioral: TAU

INTERVENTIONS:
Behavioral: SALIENCE — 3 computer-based training sessions with program "SALIENCE" per week over 3 weeks (see study description)
  Arms: TAU plus SALIENCE
Behavioral: TAU — treatment as usual, , i.e. medically supervised detoxification treatment (i.e. medical management of withdrawal symptoms, associated physical discomfort and any co-existing disorders, etc.) as well as health education and supportive therapy sessions.

SUMMARY:
This study aims to detect how the Web-based program SALIENCE affects patients with alcohol-use Disorder in terms of craving, cognitive functions and risk of relapse.

DETAILED DESCRIPTION:
In the web-based program SALIENCE ("Stop Alcohol In Everyday life - New Choices and Evaluations") the patient has to make decisions for non-alcoholic and against alcoholic drinks. Therefore there are several scenarios, which are supposed to let the patient integrate these choices into a realistic, everyday life, setting and help the patient to maintain abstinence in upcoming "high risk situations". It has been developed as an add-on therapy to increase the overall outcome.

Participating patients with alcohol-use disorder are to receive an initial screening including questionnaires and neuropsychological tests. Then the patients receive three training sessions with SALIENCE each week.

After three weeks there is another examination. After these three weeks, there is a 90 day period in which there are online follow-ups every two weeks to assess the craving and relapse of the participants. After the 90 day period there is a third examination analog to the first and the second one.

For the first 25 subjects, the follow-up and T3 will be omitted; for this collective, an interim evaluation will be performed after T2 as a pilot study, followed by optimization of the protocol if necessary. The first 25 subjects will all receive SALIENCE; a comparison with standard therapy is not planned for this collective. There will be 2 weeks between T1 and T2 in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* alcohol use disorder (DSM-5)
* inpatient or part inpatient treatment
* alcohol abstinence for at least 72 hours and maximum for three weeks
* normal or correctable eyesight
* Sufficient ability to communicate with the investigators, to answer questions in oral and written form
* "Fully Informed Consent"
* "Written Informed Consent"

Exclusion Criteria:

* Withdrawal of the declaration of consent
* severe internistic, neurological or psychiatric comorbidities
* severe withdrawal symptoms (CIWA-R > 7)
* alcohol-intoxication (> 0 ‰)
* Pharmacotherapy with psychoactive substances within the last 14 days (except Clomethiazole or Benzodiazepines within the alcohol withdrawal treatment; treatment with these medications has to be completed within last 3 days)
* Axis 1 disorder according to ICD-10 and DSM 5 (except tobacco use disorder and specific phobia within the last 12 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol craving | directly before and after each SALIENCE session (3 SALIENCE sessions per week over 3 weeks)
  Visual Analogue Scale
Change in attentional bias | directly before and after each SALIENCE session (3 SALIENCE sessions per week over 3 weeks)
  Dotprobe-Task (MacLeod, Mathews, & Tata, 1986)
Change in alcohol interference | directly before and after each SALIENCE session (3 SALIENCE sessions per week over 3 weeks)
  Alcohol Stroop Test (Brand, Leichsenring-Driessen, Beblo, Kremer, & Driessen, 2009)
Change in approach-avoidance tendencies | directly before and after each SALIENCE session (3 SALIENCE sessions per week over 3 weeks)
  Approach Avoidance Task (AAT) (R. W. Wiers et al., 2009)

SECONDARY OUTCOMES:
Relapse | 90 days after study inclusion
  time to first severe relapse

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Principal Investigator — ZI Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Weber A, Shevchenko Y, Gerhardt S, Hoffmann S, Kiefer F, Vollstadt-Klein S. Effectiveness of Reducing Craving in Alcohol Use Disorder Using a Serious Game (SALIENCE): Randomized Controlled Trial. JMIR Form Res. 2023 Nov 7;7:e42194. doi: 10.2196/42194. PMID 37934561